CLINICAL TRIAL: NCT03223363
Title: A New Birth Weight Prediction Based on Ultrasonography in Chinese Population
Brief Title: A New Birth Weight Prediction in Chinese Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: LC2016PY021
Record Dates: First submitted 2017-07-06; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Birth Weight
Keywords: Birth weight Prediction; Two-dimensional Ultrasonography; Three-dimensional Ultrasonography
MeSH Terms: conditions — Birth Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Development Group (Experimental): Development Group is used to establish the prediction model.2D and 3D ultrasonography are performed in this group. Through statistical analysis we obtain a new model.
  Interventions: Diagnostic Test: 2D and 3D ultrasonography
- Validation group (Other): Validation Group is used to confirm the efficacy of the prediction model.2D and 3D ultrasonography are performed in this group.Absolute and percentage error are calculated and compared with a common formula to confirm the accuracy of this new model.
  Interventions: Diagnostic Test: 2D and 3D ultrasonography

INTERVENTIONS:
Diagnostic Test: 2D and 3D ultrasonography — All of the examinations are performed with the same transabdominal ultrasonic transducer (RAB 2-5-D) on the same E8 (GE Medical Systems, Milwaukee, WI, USA) ultrasonic machine experienced operators. 2D ultrasonic measurements includes 5 standard fetal biometry parameters, and after routine 2D ultrasonography, the acquisition of 3D measurements are performed.

SUMMARY:
To determine the value of principal component analysis in the combined method of three-dimensional ultrasonography assessing fetal limb volume and circumference and conventional two-dimensional ultrasonography for prediction of birth weight in southern Chinese population.

DETAILED DESCRIPTION:
A prospective study was performed on single pregnant women in third trimester. Three- and two-dimensional ultrasonography for fetal biometric parameters were measured within 7 days of delivery. Stepwise linear regression were used to develop a new prediction model based on values from limb parameters and traditional measurements in development group. Estimated and actual birth weight were compared between the new model and previously published formulas on absolute error and percentage error. The accuracy of the model in predicting fetal birth weight was reassured by validation group.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria consisted of well-defined gestational age (GA), singleton pregnancy and delivery in our hospital within 7 days from the scan performed for acquisition of 2D and 3D ultrasonographic data.

Exclusion Criteria:

* The exclusion criteria were equivocal GA, multiple pregnancy, fetal severe malformation detected by prenatal ultrasonographic scans, delivery more than 7 days after the scan of 2D and 3D ultrasonography, and delivery in other institutions.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Estimated birth weight in g | 7 days within delivery
  Estimated birth weight (g) calculated by a new formula generated from ultrasonograohic parameters in development group using statistical analysis.

SECONDARY OUTCOMES:
Absolute error in g | After birth
  Absolute error (g) calculated from estimated birth weight (g) and actual birth weight (g)
Percentage error in % | After birth
  Percentage error (%) calculated from estimated birth weight (g) and actual birth weight (g)

CONTACTS AND LOCATIONS:
Overall Officials: Fang Yang, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Gynecology and Obstetrics, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Nardozza LM, Caetano AC, Zamarian AC, Mazzola JB, Silva CP, Marcal VM, Lobo TF, Peixoto AB, Araujo Junior E. Fetal growth restriction: current knowledge. Arch Gynecol Obstet. 2017 May;295(5):1061-1077. doi: 10.1007/s00404-017-4341-9. Epub 2017 Mar 11. PMID 28285426